CLINICAL TRIAL: NCT04601142
Title: Study on the Association Between the Effect of Glucocorticoid Pulse Therapy on Neuromyelitis Optica and Gene Polymorphism: a Cohort Study
Brief Title: Association Between the Effect of Glucocorticoid Pulse Therapy on Neuromyelitis Optica (NMO) and Gene Polymorphism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingTH-YLJD-202001
Record Dates: First submitted 2020-10-15; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Glucocorticoid Resistance; Gene; Neuromyelitis Optica
MeSH Terms: conditions — Glucocorticoid Receptor Deficiency; Neuromyelitis Optica | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- glucocorticoid sensitive (GS) group
  Interventions: Drug: Methylprednisolone
- glucocorticoid resistance (GR) group
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — methylprednisolone pulse therapy: 500-1000mg/d，３-５ｄ

SUMMARY:
Aims of this study are to observe the correlation between ABCB1、VDR、TBX21、NR3C1 and other gene polymorphisms and the effect of glucocorticoid shock therapy on neuromyelitis optica. Investigators plan to include patients with neuromyelitis optica who will receive glucocorticoid shock therapy prospectively. The patients are divided into glucocorticoid sensitive (GS) group and glucocorticoid resistance (GR) group according to the change of central vision after treatment. Patients' clinical data will be collected and blood samples are needed for single nucleotide polymorphism (SNP) typing test. Through statistical analysis, the data differences between GS group and GR group were compared, and the effects of clinical indexes and gene polymorphisms on the efficacy of glucocorticoid shock therapy in the treatment of neuromyelitis optica should be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of neuromyelitis optica
* Chinese Han nationality, gender is unlimited;
* Must be able to accept methylprednisolone pulse therapy

Exclusion Criteria:

* Other optic nerve diseases, such as ischemic, compressive, invasive, traumatic, toxic and nutritional metabolic, hereditary optic neuropathy;
* Visual path and central lesion on optic chiasma;
* Other eye diseases, such as anterior segment lesions, retinopathy, macular lesions, ametropia, glaucoma, etc;
* Non-organic visual impairment;
* Treated with glucocorticoid in two weeks.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New diagnosis NMO patients who plan to receive methylprednisolone pulse therapy.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the change of best corrected visual acuity (BCVA) | 3 day after the treatment of methylprednisolone pulse therapy
  Test BCVA before and after the treatment of methylprednisolone pulse therapy, and calculate the change value

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided